CLINICAL TRIAL: NCT02869906
Title: Instantaneous Wave-Free Ratio and Fractional Flow Reserve for the Assessment of Non Culprit Lesions in Patients With ST-segment Elevation Myocardial Infarction
Acronym: WAVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Principal Investigator, Carmine Musto, MD PhD, Azienda Ospedaliera San Camillo Forlanini
Other Study IDs: 1510/2016 CE Lazio 1
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FFR and iFR: The investigators compare FFR and iFR values in the acute phase of STEMI and in the subacute phase, 5-7 days after STEMI.
  Interventions: Other: FFR and iFR

INTERVENTIONS:
Other: FFR and iFR — The investigators aimed to assess the reliability of the instantaneous wave-free ratio (iFR) and fractional flow reserve (FFR) measurements in non-culprit coronary lesions during the acute and subacute phase of ST-segment elevation myocardial infarction (STEMI).

SUMMARY:
Functional assessment of non-culprit lesions during percutaneous coronary intervention (PCI) in patients with acute coronary syndrome could improve risk stratification and shorten the duration of hospital stay by decreasing the need for additional non-invasive stress testing to detect residual myocardial ischemia. The investigators aimed to assess the reliability of the instantaneous wave-free ratio (iFR) and fractional flow reserve (FFR) measurements in non-culprit coronary lesions during the acute and subacute phase of ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
BACKGROUND: Approximately 30% of patients who present with ST elevation myocardial infarction have multivessel coronary artery disease on angiography. Whether percutaneous coronary intervention (PCI) should be limited to the culprit lesion only or applied to all angiographically critical non-culprit lesions is still debatable. The FAME 2 study has shown that Fractional Flow Reserve (FFR)-guided PCI, with adenosine infusion, reduces the MACE compared to medical therapy alone. In fact, according to the recent ESC clinical guidelines, FFR guided PCI is in class I, evidence level A. Previous studies, have confirmed that FFR values of non-culprit coronary lesions in STEMI patients provided similar values in the acute phase compared to the subacute phase, 5-7 days after primary PCI. Consequently, it is possible to assess angiographically borderline non-culprit lesions during the acute phase and hence risk stratify STEMI patients, thus reducing the duration of hospital stay by decreasing the need for additional non-invasive stress testing to detect residual myocardial ischemia. However, the assessment of angiographically borderline lesions using FFR has its own limitations related to the use of adenosine, which increases the risk of bradyarrhythmias and high degree atrioventricular block, especially in the acute phase. This would make functional assessment of the non-culprit lesions not always possible during the acute phase.

Recently, a new functional algorithm, called "instantaneous wave-free ratio" (iFR) has been introduced. Similar to FFR, it gives a functional assessment of coronary lesions by measuring the trans-stenotic gradient during ventricular diastole, where intramyocardial resistance is minimal and constant. This phase has been shown to be comparable to the maximum hyperemic state of FFR assessment.

The measurement of iFR during the acute phase of STEMI has not yet been evaluated.

AIM: The aim of this study is to assess the reliability of the instantaneous wave-free ratio (iFR) and fractional flow reserve (FFR) measurements in non-culprit coronary lesions during the acute and subacute phase of ST-segment elevation myocardial infarction (STEMI).

METHOD: Patients undergoing primary PCI for STEMI and presenting with multivessel coronary disease (at least one ≥ 50% diameter stenosis in a non-infarct-related coronary artery) were enrolled in a prospective observational registry. Coronary lesions were evaluated with both iFR and FFR immediately after primary PCI (acute phase) and 7 ± 3 days later (subacute phase).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary PCI for STEMI and presenting with multivessel coronary disease (at least one ≥ 50% diameter stenosis in a non-infarct-related coronary artery) were enrolled.

Exclusion Criteria:

* severe left ventricular dysfunction (Ejection Fraction <30%).
* Heart Failure
* Previous STEMI
* Severe sinus bradycardia
* Past medical history of Asthma
* TIMI flow 1,2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary PCI for STEMI and presenting with multivessel coronary disease (at least one ≥ 50% diameter stenosis in a non-infarct-related coronary artery).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of iFR and FFR values in the non culprit lesion during STEMI in the acute and subacute phase. | 5-7 days
  Comparison of iFR and FFR values for evaluating the functional significance of non-culprit coronary lesions in patients with STEMI, both during primary PCI and during staged procedures,

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Musto, PhD, Principal Investigator — Ospedale San Camillo
Locations (1):
- Ospedale San Camillo, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided